CLINICAL TRIAL: NCT04875780
Title: Effects of a Smartphone-based Weight Loss Programme Targeting Chinese Overweight Adults With Pre-diabetes: A Randomized Controlled Trial
Brief Title: A Smartphone-based Intervention for Diabetes Prevention in Overweight Chinese Adults With Pre-diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Mandy M. Ho, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HMRF03180248
Record Dates: First submitted 2021-05-01; First posted 2021-05-06 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Pre-diabetes
Keywords: Diabetes prevention; Pre-diabetes; Weight loss; Cardio-metabolic risk; Obesity; Lifestyle intervention; Smartphone-based
MeSH Terms: conditions — Glucose Intolerance; Weight Loss; Obesity

STUDY DESIGN:
Intervention Model Description: It is a 12-month 3-arm randomised controlled trial, RCT (the digital diabetes prevention app group, the digital weight loss tracking app group, and the wait-list usual care group). The digital diabetes prevention app group will receive these intervention components: web-based diabetes prevention curriculum, virtual social group support, goal setting and self-monitoring via the smartphone app. The digital weight loss tracking group will receive digital tracking of weight loss, diet and physical activity and virtual social support group function (mimicking the publically available weight loss apps), but without the web-based diabetes prevention curriculum.
  The wait-list usual care group will receive usual care in the form of an annual review and blood test, together with general lifestyle advice at our NGO collaborator's (UCN) community clinics.
Who Masked: Outcomes Assessor
Masking Description: All outcome assessors will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digital diabetes prevention app intervention (Experimental): Participants will receive web-based diabetes prevention curriculum, virtual social group support and digital tracking via the smartphone app.
  Interventions: Behavioral: Digital diabetes prevention app intervention
- Digital weight loss tracking app intervention (Active Comparator): Participants will receive the same intervention as the digital diabetes prevention curriculum app group except the web-based diabetes prevention curriculum.
  Interventions: Behavioral: Digital weight loss tracking app intervention
- Wait-list control (usual care) (Other): Participants will receive usual care in the form of an annual review and blood test, together with general lifestyle advice.
  Interventions: Behavioral: Wait-list control (usual care)

INTERVENTIONS:
Behavioral: Digital diabetes prevention app intervention — 16-week core program consisting of 16 online weekly interactive lessons on diet and physical activity for weight loss. After the completion of the core program, participant can proceed to the 36-week post-core phase. The post-core program provides 8 monthly lessons focusing on maintaining lifestyle habits and weight loss.
  Participants will be guided to use the smartphone app for goal setting and self-monitoring of diet, physical activity and weight loss.
  Participants will be demographically matched into online groups of 10-12 persons. Online group discussion board will be set up for participants to discuss goals, share progress and provide supports to each other.
  Other Names: Web-based diabetes prevention curriculum; Goal setting and self-monitoring; Virtual social support group
  Arms: Digital diabetes prevention app intervention
Behavioral: Digital weight loss tracking app intervention — All participants will be provided the same smartphone app as the intervention group for goal setting and self-monitoring of diet, physical activity and weight loss.
  Participants will be demographically matched into online groups of 10-12 person. Online group discussion board will be set up for participants to discuss goals, share progress and provide supports to each other.
  Other Names: Goal setting and self-monitoring; Virtual social support group
  Arms: Digital weight loss tracking app intervention
Behavioral: Wait-list control (usual care) — Participants in the control group will be invited to have an annual review and blood test at baseline, 4 and 12 months and received general lifestyle advices from a registered nurse at a community clinic.
  Arms: Wait-list control (usual care)

SUMMARY:
Type 2 diabetes (T2DM) is a serious chronic condition and one of the world's fastest growing health problems. The onset of T2DM is gradual, with most individuals progressing through a state of pre-diabetes, which provides an important window of opportunity for the prevention of T2DM and its complications. This project aims to translate the evidence-based diabetes prevention strategies into community setting and utilize mobile health technology to reduce diabetes risks in Hong Kong.

DETAILED DESCRIPTION:
Type 2 diabetes (T2DM) is a major global health issue and the cost to community is high and escalating. The Asia-Pacific region carries a high disease burden, with more than 60% of the global diabetic population living in Asian region. The onset of T2DM is gradual, with most individuals progressing through a state of pre-diabetes. A National Survey conducted in China in 2010 revealed that 50.1% of people aged 18 or older have pre-diabetes. People with pre-diabetes, defined as having impaired fasting glucose (IFG), impaired glucose tolerance (IGT) or elevated glycated haemoglobulin (HbA1C) , are at increased risk of developing T2DM and its associated complications, such as heart diseases and retinopathy, which can develop even in the absence of progression to overt T2DM. Hence, it is essential that people with pre-diabetes are targeted for early intervention to prevent T2DM and related complications.

Obesity is a major risk factor for developing T2DM. International trials demonstrate that lifestyle interventions (which includes diet, physical activity and behavioural modification components) targeting at least 5% weight loss in individuals with pre-diabetes can reduce 3-year diabetes incidence by 58%. Growing evidence suggests that smartphones may be a promising platform for delivery of behavioural lifestyle intervention to achieve weight loss.

This project aims to translate the evidence-based diabetes prevention strategies into community setting and utilize mobile health technology to reduce diabetes risks in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 40 - 60 years old
* Overweight (BMI ≥ 23kg/m2) or obese (BMI ≥ 25 kg/m2)
* With at least one blood test result showing IGT (7.8-11.0 mmol/L after a two-hour glucose tolerance test), IFG (fasting glucose 5.6 - 6.9 mmol/L) or impaired HbA1c 5.7% - 6.4%
* Owns a smartphone
* Able to read Chinese and speak Cantonese.

Exclusion Criteria:

* With current or clinical history of T2DM, or with co-morbid conditions that may limit participation in the study, such as recent history of an acute cardiovascular event, uncontrolled hypertension, cancer or major psychiatric or cognitive problems
* Already participating in a weight loss programme
* Receiving drug treatment for pre-diabetes or long-term use of medicines known to influence glucose metabolism (e.g. corticosteroids)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 282 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Percent weight change | % weight change at 4 and 12 months from baseline
  % weight change from baseline

SECONDARY OUTCOMES:
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Changes of insulin sensitivity at 12-months from baseline
  Estimated from fasting insulin and fasting glucose, [fasting insulin (uU/mL)*fasting glucose(mmol/L)]/22.5
Fasting insulin | Changes of fasting insulin to 12-months from baseline
  Fasting insulin in mU/L
Fasting blood glucose (FG) | Changes of FG at 12-months from baseline
  Fasting blood glucose in mmol/L > 8 hours of fasting
Haemoglobin A1C (HbA1C) | Changes of HbA1c at 4 and 12-months from baseline
  HbA1c in %
Systolic and diastolic blood pressure (SBP, DBP) | Changes of SBP and DBP to 4 and 12-months from baseline
  in mmHg measured by automatic BP monitor
Blood lipid profile | Changesof blood lipid at 12-months from baseline
  fasting blood for total cholesterol, HDL, LDL and triglycerides, all in mmol/L
2hr post OGTT glucose (2hr PP) | Changes of 2hr PP at 12-months from baseline
  Blood glucose in mmol/L 2 hours after OGTT
Physical activity as assessed by IPAQ | Change in levels of physical activity from baseline to 4 and 12-months
  International physical activity questionnaire short form (IPAQ, Chinese version). A validated 6-item questionnaire to assess the frequency and duration of vigorous intensity activity, moderate intensity activity, and walking. The questionnaire will be scored using established methods (www.ipaq.ki.se). Data will be summarized to report physical activity in categories:
  1. High-active group
     * Vigorous-intensity activity on ≥ 3 days and accumulating ≥1500 MET-minutes/week OR
     * ≥7 days of any combination of walking, moderate-intensity or vigorous intensity activities achieving ≥3000 MET-minutes/week
  2. Moderate-active group
     * ≥3 days of vigorous activity of ≥20 minutes/day OR
     * ≥5 days of moderate-intensity activity or walking of ≥30 minutes/day OR
     * ≥5 days of any combination of walking, moderate-intensity or vigorous intensity activities achieving ≥600 MET-min/week.
  3. Low-active/inactive group Individuals who do not meet criteria for high- and moderate-active
Dietary intake as assessed by 24-hour recall | Changes in dietary intake from baseline to 4 and 12-months
  24-hour food recall
Health-related quality of life (HRQOL) as assessed by SF12 | Changes in HRQOL from baseline to 4 and 12-months
  12-item Short Form Survey (SF12 Chinese version). It is a validated scale which provides two summary measures.
  Physical and Mental Health Composite Scores (PCS & MCS) will be computed using the scores of 12 questions and range from 0 to 100. Higher scores represent better health.
Central obesity | Changes of waist circumference at 12-months from baseline
  Waist circumference in cm
Percentage body fat as assessed by BIA | Changes of body fat at 12-months from baseline
  Bioelectrical impedance analysis measuring body fat in %
Smartphone apps user engagement | At 12-months follow-up
  User's overall login frequency and duration to the app and login frequency and duration to each module, as well as the frequency of participation in the group sharing and discussion. Usage data will be obtained from the apps administrative portal.
User feedback as assessed by an online exit questionnaire | At 12-months follow-up
  An online exit questionnaire will be administered to participants in the intervention group at 12 months.

OTHER OUTCOMES:
Diabetes incidence | At 12-months follow-up
  Oral glucose tolerance test (OGTT) in mmol/L measured 2 hours after 75g oral glucose intake post overnight fast. Diabetes is defined as FG≥7.0mmol/L or 2hr post OGTT ≥ 11.1mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mandy Ho, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] American Diabetes Association. (2) Classification and diagnosis of diabetes. Diabetes Care. 2015 Jan;38 Suppl:S8-S16. doi: 10.2337/dc15-S005. No abstract available. PMID 25537714
- [Background] Guariguata L, Whiting DR, Hambleton I, Beagley J, Linnenkamp U, Shaw JE. Global estimates of diabetes prevalence for 2013 and projections for 2035. Diabetes Res Clin Pract. 2014 Feb;103(2):137-49. doi: 10.1016/j.diabres.2013.11.002. Epub 2013 Dec 1. PMID 24630390
- [Background] Mirasol R, Thai AC, Salahuddin AA, Tan K, Deerochanawong C, Mohamed M, Saraswati MR, Sethi BK, Shah S, Soetedjo NN, Suraamornkul S, Tan R, Uddin F. A Consensus of Key Opinion Leaders on the Management of Pre-diabetes in the Asia-Pacific Region. J ASEAN Fed Endocr Soc. 2017;32(1):6-12. doi: 10.15605/jafes.032.01.02. Epub 2017 May 5. PMID 33442078
- [Background] Yoon KH, Lee JH, Kim JW, Cho JH, Choi YH, Ko SH, Zimmet P, Son HY. Epidemic obesity and type 2 diabetes in Asia. Lancet. 2006 Nov 11;368(9548):1681-8. doi: 10.1016/S0140-6736(06)69703-1. PMID 17098087
- [Background] Chan JC, Zhang Y, Ning G. Diabetes in China: a societal solution for a personal challenge. Lancet Diabetes Endocrinol. 2014 Dec;2(12):969-79. doi: 10.1016/S2213-8587(14)70144-5. Epub 2014 Sep 10. PMID 25218728
- [Background] Singleton JR, Smith AG, Russell JW, Feldman EL. Microvascular complications of impaired glucose tolerance. Diabetes. 2003 Dec;52(12):2867-73. doi: 10.2337/diabetes.52.12.2867. PMID 14633845
- [Background] Levitan EB, Song Y, Ford ES, Liu S. Is nondiabetic hyperglycemia a risk factor for cardiovascular disease? A meta-analysis of prospective studies. Arch Intern Med. 2004 Oct 25;164(19):2147-55. doi: 10.1001/archinte.164.19.2147. PMID 15505129
- [Background] Nathan DM, Davidson MB, DeFronzo RA, Heine RJ, Henry RR, Pratley R, Zinman B; American Diabetes Association. Impaired fasting glucose and impaired glucose tolerance: implications for care. Diabetes Care. 2007 Mar;30(3):753-9. doi: 10.2337/dc07-9920. No abstract available. PMID 17327355
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Gong Q, Gregg EW, Wang J, An Y, Zhang P, Yang W, Li H, Li H, Jiang Y, Shuai Y, Zhang B, Zhang J, Gerzoff RB, Roglic G, Hu Y, Li G, Bennett PH. Long-term effects of a randomised trial of a 6-year lifestyle intervention in impaired glucose tolerance on diabetes-related microvascular complications: the China Da Qing Diabetes Prevention Outcome Study. Diabetologia. 2011 Feb;54(2):300-7. doi: 10.1007/s00125-010-1948-9. Epub 2010 Nov 3. PMID 21046360
- [Background] Lindstrom J, Peltonen M, Eriksson JG, Ilanne-Parikka P, Aunola S, Keinanen-Kiukaanniemi S, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study (DPS). Improved lifestyle and decreased diabetes risk over 13 years: long-term follow-up of the randomised Finnish Diabetes Prevention Study (DPS). Diabetologia. 2013 Feb;56(2):284-93. doi: 10.1007/s00125-012-2752-5. Epub 2012 Oct 24. PMID 23093136
- [Background] Schoeppe S, Alley S, Van Lippevelde W, Bray NA, Williams SL, Duncan MJ, Vandelanotte C. Efficacy of interventions that use apps to improve diet, physical activity and sedentary behaviour: a systematic review. Int J Behav Nutr Phys Act. 2016 Dec 7;13(1):127. doi: 10.1186/s12966-016-0454-y. PMID 27927218
- [Background] Sepah SC, Jiang L, Ellis RJ, McDermott K, Peters AL. Engagement and outcomes in a digital Diabetes Prevention Program: 3-year update. BMJ Open Diabetes Res Care. 2017 Sep 7;5(1):e000422. doi: 10.1136/bmjdrc-2017-000422. eCollection 2017. PMID 28948027
- [Background] Khokhar B, Jones J, Ronksley PE, Armstrong MJ, Caird J, Rabi D. Effectiveness of mobile electronic devices in weight loss among overweight and obese populations: a systematic review and meta-analysis. BMC Obes. 2014 Oct 14;1:22. doi: 10.1186/s40608-014-0022-4. eCollection 2014. PMID 26217509
- [Background] Azar KM, Lesser LI, Laing BY, Stephens J, Aurora MS, Burke LE, Palaniappan LP. Mobile applications for weight management: theory-based content analysis. Am J Prev Med. 2013 Nov;45(5):583-9. doi: 10.1016/j.amepre.2013.07.005. PMID 24139771
- [Background] Semper HM, Povey R, Clark-Carter D. A systematic review of the effectiveness of smartphone applications that encourage dietary self-regulatory strategies for weight loss in overweight and obese adults. Obes Rev. 2016 Sep;17(9):895-906. doi: 10.1111/obr.12428. Epub 2016 May 18. PMID 27192162
- [Background] Michie S, Ashford S, Sniehotta FF, Dombrowski SU, Bishop A, French DP. A refined taxonomy of behaviour change techniques to help people change their physical activity and healthy eating behaviours: the CALO-RE taxonomy. Psychol Health. 2011 Nov;26(11):1479-98. doi: 10.1080/08870446.2010.540664. Epub 2011 Jun 28. PMID 21678185
- [Background] World Health Organization. Definition and diagnosis of diabetes mellitus and intermediate hyperglycemia: report of a WHO/IDF consultation. Geneva: 2006.